CLINICAL TRIAL: NCT04405557
Title: Study on the Application of ctDNA in a Population at High-risk for Common Malignant Tumor
Brief Title: The PREDICT Study: Prospective Early Detection In a Population at High-risk for Common Malignant Tumor
Status: Active, not recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT
Record Dates: First submitted 2020-05-09; First posted 2020-05-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Early Detection of Cancer
Keywords: Pan-cancer; cancer screening; ctDNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a observational, multicenter study, monitoring the circulating tumor DNA (ctDNA) in people who is at risk of cancers，assessing the sensitivity and specificity of ctDNA detection in early screening of pan-carcinoma.

DETAILED DESCRIPTION:
2000 patients with positive tumor protein markers or cancer screening were recruited. All patients were tested for ctDNA at enrollment and followed up at 6 months and 1 year. The study was completed at the time of cancer diagnosis or the longest follow-up time (1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged at or over 45 years old.
2. Patients who with one or more of the following situations:

   1. In AFP (>20UG/L), CA125 (>70U/ml), CEA (>7ng/ml) and CA199 (>60U/ml), more than one item was abnormal for two consecutive times within one month.
   2. Patients with viral hepatitis (Hepatitis B / C surface antigen positive with liver function damage.
   3. Patients with liver nodules detected by ultrasound and hemangioma excluded.
   4. Patients with compensated cirrhosis.
   5. CA125>35U/ml and HE4 was abnormal (the reference value of HE4 in premenopausal and postmenopausal women was 68.96 pmol/L and 114.90 pmol/L respectively).
   6. Patients with ovarian masses found by ultrasonography (premenopausal > 5cm, postmenopausal > 3.5cm).
   7. Patients with pancreatic space-occupying found by ultrasonography.
   8. Patients with BI-RADS grade 4 or above by ultrasound or mammography.
   9. CA125>35U/ml and BI-RADS above grade 3 by ultrasound or mammography.
   10. CA153>25U/ml and BI-RADS above grade 3 by ultrasound or mammography.
   11. Family genetic history of breast cancer and ovarian cancer, and BI-RADS above grade 3 by ultrasound or mammography.
   12. Patients with a positive fecal occult blood test and haemorrhoids excluded
   13. Patients with a positive fecal occult blood test and positive CEA
   14. More than 2 items were abnormal in PGI, PGR and G-17 (criteria: PGI≤70 UG/L, PGR≤7.0, G-17≤1 pmol/L or G-17≥15 pmol/L).
3. Ability to collect specimens from each time point and provide corresponding clinical information.
4. Understand the research plan and voluntarily participate in the study, sign the informed consent form.

Exclusion Criteria:

1. Patients with previous or present cancer.
2. Patients with serious diseases, especially those with a survival period of less than 3 years.
3. Patients with factors that affect the diagnosis of the disease (such as MRI related cardiac pacemakers, ferromagnetic implants, etc.).
4. Patients with a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
5. Women who are pregnant or preparing for pregnancy.
6. Patients who voluntarily withdraw for any reason.
7. Patients who cannot complete the research plan

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with positive tumor protein marker or cancer screening.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of ctDNA for early detection in cancer high-risk population. | 1 year
  To evaluate the sensitivity, specificity and positive predictive value of ctDNA for screening in high-risk population. Including the following six types of cancer: hepatocellular carcinoma, pancreatic cancer, ovarian cancer, breast cancer, colorectal cancer and gastric cancer.

SECONDARY OUTCOMES:
Window period from ctDNA positive to cancer diagnosis. | 1 year
  To evaluate the time from ctDNA positive to cancer diagnosis for patients diagnosed with cancer during the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zeng, MD, Principal Investigator — Chinese PLA General Hospital
Locations (8):
- China (8):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan